CLINICAL TRIAL: NCT02887547
Title: Biomarkers Expression in Gingival Crevicular Fluid and Accelerated Tooth Movement
Brief Title: Biological Markers Evaluation of Accelerated Tooth Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, LIANA FATTORI ABATI, MS, PhD, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Fattori2
Record Dates: First submitted 2015-12-20; First posted 2016-09-02 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Cytokine Measurements; Orthodontic Space Closure; Tooth Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group, with traditional orthodontic mechanics for anterior retraction. Crevicular fluid will be collected during anterior retraction mechanics to identified biomarkers in the inflammatory process
- Acceleration (Experimental): Group with micro-osteoperforation for accelerated tooth movement during anterior retraction, Crevicular fluid will be collected during anterior retraction mechanics to identified biomarkers in the inflammatory process
  Interventions: Procedure: micro-osteoperforation

INTERVENTIONS:
Procedure: micro-osteoperforation
  Other Names: accelerated tooth movement
  Arms: Acceleration

SUMMARY:
Gingival Crevicular Fluid samples will be collected using periopapers after accelerated tooth movement technique, results will be assessed with biomarkers levels done using ELISA Assays

DETAILED DESCRIPTION:
For this prospective study, 22 individuals were selected, with skeletal discrepancies randomly divided into two groups: 1 - accelerated tooth movement technique (ATMT) and 2 - Control.

Orthodontic records done in two times, initial and preoperative; Gingival Crevicular Fluid samples will be collected using periopapers in 7 times (1, 2, 7, 14, 28 days and after space closure- end of orthodontic treatment movement activation).

Flapless cortical perforations will be made in ATMT Group after dental extraction. Surgical protocol will be flapless to preserve periodontal health.

After extraction space closure, results will be assessed by clinical effects with biological markers levels:

CCL3/MIP-1 alpha, CCL5/RANTES, CXCL8/IL8, IL-1 alpha, IL-1 beta, IL6, TNF-alpha, TRANCE/RANK L, OCN OPG IL-10 VEGF TGF-ℬ

Those biomarkers levels will be performed using ELISA Assays. After collecting data, the results will be statistically analyzed using Shapiro-Wilk and, posteriorly, T-student or Wilcoxon.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ages 18-40 years old, in good general health, with adult complete dentition, regardless of presence of third molars.
* Indication for orthognathic surgery
* Tooth extraction indication for orthodontic treatment
* Do not smoke
* Periodontal and teeth healthy
* Do not use bisphosphonates or corticosteroids

Exclusion Criteria:

* Surgically assisted rapid palatal expansion indication
* Cleft lip and palate
* Craniofacial syndrome
* Mental disorder
* Metabolic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Cytokines ad Chemokines Detection Assay | 8 months
  Measure the different levels of listed cytokines and chemokines after starting the anterior retraction
Bone remodeling markers in GCF samples | 8 monnths
  Measure the different levels of resorption biomarkers and bone formation after starting the anterior retraction

CONTACTS AND LOCATIONS:
Overall Officials: Liana Fattori, MS PhD, Principal Investigator — Phd candidate; Jose Rino Neto, Study Chair — University of Sao Paulo